CLINICAL TRIAL: NCT06617247
Title: Effects of Cannabidiol on Burnout Syndrome and Empathy of Paid and Unpaid Caregivers of Older Adults
Brief Title: Effects of Cannabidiol on Burnout Syndrome and Empathy of Caregivers of Older Adults
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Madson Alan Maximiano-Barreto, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 79253324.5.0000.5440
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Burnout Syndrome
Keywords: cannabidiol; caregivers; empathy; Burnout syndrome
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, double-blind, placebo-controlled two-arm clinical trial to achieve the main objective of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention 2: Placebo (Experimental): In this group, the subjects will receive placebo intervention. For blinding purposes, caregivers in this group will use the vehicle of oral CBD 300mg (150mg twice
  Interventions: Drug: Intervention 2: Placebo
- Intervention1: Cannabidiol (Experimental): The caregivers randomized for this intervention will use oral CBD 300 mg (i.e., 150mg, twice daily) for four weeks. The substance will be provided free of charge by the company Ease Labs, and will be administered in capsules to promote blinding. This posology was based on the study, in which CBD in this dosage and form of presentation proved to be safe and effective in reducing indicators of burnout in frontline health professionals from COVID-19. The safety of CBD use has also been reported in previous studies conducted with humans. Side effects from CBD use are rare, including mild and tolerable symptoms (e.g., dizziness, drowsiness, fatigue, lethargy, nausea, headache, fever, and sensory changes).
  Interventions: Drug: Intervention1: Cannabidiol

INTERVENTIONS:
Drug: Intervention1: Cannabidiol — Os cuidadores randomizados para esta intervenção usarão CBD oral 300 mg (ou seja, 150 mg, duas vezes ao dia) por quatro semanas. A substância será fornecida gratuitamente pela empresa Ease Labs e será administrada em cápsulas para promover o cegamento. Esta posologia foi baseada no estudo, no qual o CBD nesta dosagem e forma de apresentação provou ser seguro e eficaz na redução de indicadores de burnout em profissionais de saúde da linha de frente da COVID-19. A segurança do uso do CBD também foi relatada em estudos anteriores conduzidos com humanos. Os efeitos colaterais do uso do CBD são raros, incluindo sintomas leves e toleráveis (por exemplo, tontura, sonolência, fadiga, letargia, náusea, dor de cabeça, febre e alterações sensoriais).
  Arms: Intervention1: Cannabidiol
Drug: Intervention 2: Placebo — In this group, the subjects will receive placebo intervention. For blinding purposes, caregivers in this group will use the vehicle of oral CBD 300mg (
  Arms: Intervention 2: Placebo

SUMMARY:
Burnout syndrome is an occupational disease that has affected health care providers, for example, caregivers of older adults. This syndrome negatively affects physical and psychological health, which may reflect on the mental health of the caregiver and the care provided to the older adults. Interventions have been developed to minimize the impacts of burnout. Thus, this study has two main objectives: 1) to identify the effect of cannabidiol on indicators of burnout and empathy of caregivers of older people with functional dependence for activities of daily living; 2) identify possible associations between burnout indicators, empathy levels and their domains, and quality of care. This is a two-phase study (i.e., Phase 1: cross-sectional; Phase 2: clinical trial). In Phase 1, caregivers will answer questionnaires developed by researchers for sociodemographic characterization, care and satisfaction of care. In addition, they will complete instruments to assess the functional dependence of the older people - EIAVD, depressive symptoms - PHQ-9, social support - EAS, Burnout syndrome - MBI and Empathy - EMRI and MET. In Phase 2, caregivers will be randomized to cannabidiol or placebo intervention. Caregivers with number 0 will be allocated to the intervention using cannabidiol (300mg - divided into two times a day) and those drawn with number 1 will be allocated to the placebo group. Both interventions will be performed for four weeks. Caregivers will fill in the MBI, EMRI, MET, NPI and QAO instruments before and after the intervention. UKU-SERS will also be applied to evaluate side effects, IECC to assess the impact of intervention on care and CGI to assess severity and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Total score 4 in the IEAVD
* Score on the emotional exhaustion subscale of MBI 9 and/or depersonalization 6 and/or; professional achievement 10
* Low level of empathy in the EMRI scale (i.e., total score 71)
* In addition, they should have a score of 10 on the PHQ-9, indicating absence of expressive depressive symptoms

Exclusion Criteria:

* Not have the availability to participate in this phase of the research will be excluded
* Who have ceased to exercise the position of carer of a person aged 60 years or more
* Who no longer perform minimum workload of six hours daily and
* Not complete the protocol of the intervention received.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Interpersonal Reactivity Index - IRI | From enrollment to the end of treatment at 4 weeks
  IRIis a self-assessment instrument, developed for the purpose of multidimensional empathy evaluation, and will be used the version adapted and translated into Brazilian Portuguese. The Brazilian version of IRI evaluates dimensions (i.e., perspective taking, empathic consideration and personal anguish) and is composed by 21 questions (seven items to evaluate cognitive domain and 14 for evaluation of affective domain) with answers from one (low empathy) to five (high empathy) and the higher your score, the higher the level of empathy.
Multifaceted Empathy Test - MET | From enrollment to the end of treatment at 4 weeks
  The MET is a computerized instrument that allows to evaluate separately the affective and cognitive domains of empathy. The application of this instrument is performed on a computer and consists of photographs that depict people in different emotional situations (i.e., positive and negative). To assess cognitive empathy, subjects must infer the mental states of individuals shown in the images by selecting one of four descriptors of mental state (e.g., proud, joy, happy, relieved). To assess affective empathy, subjects evaluate their level of empathic concern for the individuals shown in the images on a likert scale from 1 (no little) to 9 (extremely) points. The translated version will be used and adapted to the Brazilian context.
Kliniske Undersøgelser Side Effect Rating Scale - UKU-SERS | From enrollment to the end of treatment at 4 weeks
  The safety and tolerability of the use of cannabidiol will be evaluated by UKU-SERS. Developed to evaluate the side effects and psychodrugs of the clinical research committee of the Scandinavian society of psychopharmacology. It is a self-applicable instrument that evaluates the severity of symptoms and perception of side effects in relation to four dimensions (i.e., psychiatric, neurological, autonomic and others) in 48 items with a likert response ranging from 0 to 3 and a total score ranging from 0 to 144.
  Acceptance will be evaluated by the percentage of participants who dropped out for other reasons not related to tolerability. This instrument in particular, will be applied by means of connection (i.e., weekly) and assisted at the end of the intervention, given a possible difficulty in understanding technical terms, the researcher will read, explain the criterion and score the instrument together with volunteer. This instrument will be used as a primary
Maslach's Burnout Inventory - MBI | From enrollment to the end of treatment at 4 weeks
  The objective of the scale is to evaluate the presence of Burnout Syndrome as a consequence of overload caused by chronic stress factors experienced in the work environment. This is an inventory that evaluates three main dimensions (emotional exhaustion, depersonalization and professional achievement) composed of 9 items scored on a likert scale: for each of the questions are assigned increasing intensity degree 0 (never) to 6 (daily). The translated and validated version for the Brazilian context was performed and this will be used in this study. The following scores were adopted for each subscale: emotional exhaustion 9; depersonalization 6 and; professional achievement 10.

SECONDARY OUTCOMES:
Questionnaire of assistance offered - QAO | From enrollment to the end of treatment at 4 weeks
  An instrument developed by researchers to evaluate the assistance provided by caregivers of elderly people. It consists of 10 items, scored on a likert scale (0 (very dissatisfied) to 4 (very satisfied)), to be answered by the caregiver. The score of this instrument will have a range between 0 and 40 and the higher the score, the better the assistance provided to the person receiving care (i.e., elderly).
Neuropsychiatric Inventory - NPI | From enrollment to the end of treatment at 4 weeks
  The NPI is an inventory developed that aims to evaluate the frequency and severity of neuropsychiatric symptoms. This instrument presents scores for the severity of symptoms ranging from 1 to 3 (1 = mild; 2 = moderate; 3 = severe) and frequency from 0 to 4 (0 = not disturbing; 5 = extreme). It is a likert type instrument composed of 12 items where its total score (sum of the frequency x intensity of the items) varies from 0 to 120 points. The translated version will be used and adapted to Brazilian Portuguese. This instrument is applied to the caregiver and evaluates neuropsychiatric symptoms of care recipients and will be a secondary outcome of the study, with the objective of evaluating the impact of the intervention on care recipients (i.e., older people). This instrument will be evaluated before and after the intervention in Phase 2.
Impact of possible side effects associated with CBD use | From enrollment to the end of treatment at 4 weeks
  This questionnaire was developed with the objective of evaluating the impact of some possible side effects associated with the use of CBD in the provision of care to the elderly. The study that evaluated the effect of CBD on Burnout syndrome in health professionals who worked on the front line of COVID-19, which identified the following side effects: fatigue, increased appetite, weight gain, diarrhea and lethargy, effects also observed in other studies. Therefore, this questionnaire was included in the study using adapted questions of specific measures for headache (HIT-6 TM), sleep (PSQI-BR), gastrointestinal symptoms (GSRS) and lightheadedness (DHI). The questionnaire is composed of six questions scored on a dichotomous scale (Yes/No).
Global Clinical Printing - CGI | From enrollment to the end of treatment at 4 weeks
  The CGI is a simple and fast application instrument, validated for the Brazilian context, used to evaluate the severity of symptoms and response to treatment in patients with mental disorders (e.g., depression). This instrument is used in naturalistic studies and clinical practice. It is a scale of three items evaluated by the observer, which evaluates five dimensions (i.e., positive, negative, cognitive, depressive and global symptoms) in a score ranging from 1 (normal) to 7 (highest level of severity). CGI has proven to be a robust measure of efficacy in many clinical trials of drugs and is easy and quick to administer.

OTHER OUTCOMES:
Patient Health Questionnaire - PHQ-9 | From enrollment to the end of treatment at 4 weeks
  PHQ-9 is based on the criteria for tracing episodes of depression according to the Diagnostic and Statistical Manual of Mental Disorders - DSM. It is an instrument with nine items that allows to investigate in the previous two weeks depressed mood, anhedonia, sleep, tiredness/lack of energy, change/ lack of appetite, uselessness/guilt, concentration and/or slowness/restlessness and suicidal thoughts. Their responses are scored on a likert scale from zero to three, the total score goes from 0 to 27 and the higher the score, more depressive symptoms. This instrument will be used for sample characterization in Phase 1 and will be used as a control variable in Phase 2.
Independence Scale in Daily Life Activities - ESDLA | From enrollment to the end of treatment at 4 weeks
  ESDLA was developed to assess the dependence of people (e.g., elderly people) on basic activities of daily living such as feeding, sphincter control, transfer, hygiene and fitness for dressing and bathing. It was translated and validated for the Brazilian context. This instrument is composed of six items, with likert type responses (0 to 2 points: very dependent; 3 to 4 points: moderately dependent; and 5 to 6 points: independent). This instrument used for inclusion and/or exclusion of subjects will be answered by the participants in the study regarding the level of independence of the person cared for. For the purposes of this study, the cut-off grade greater than or equal to four will be adopted, indicating the degree of dependence on activities of daily living.
Sociodemographic and care questionnaire | From enrollment to the end of treatment at 4 weeks
  This questionnaire was developed by the researchers with the objective of characterizing the sample as to variables: age (in years), sex (male/female), marital status (with partner/without partner), education level (in years). It will also make it possible to characterize the profile of caregivers: paid or not, time (in months), days of the week and hours of care.

CONTACTS AND LOCATIONS:
Locations (1):
- University os São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Following ethical recommendations and guaranteed the security of anonymity of IPD.